CLINICAL TRIAL: NCT06077734
Title: In Vitro Quality Assessment of Myogenic Stem Cells in Multiple Patient Groups With Confirmed Skeletal Muscle Atrophy to Study Their Potential for Autologous Stem Cell Therapy
Brief Title: Muscle Stem Cell Quality in Atrophy
Acronym: ATROMAB
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL 81090.068.22
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Muscle Weakness; Atrophy, Muscle; Cachexia; Sarcopenia; Stem Cell Transplantation; Mesenchymal Stem Cells
MeSH Terms: conditions — Muscle Weakness; Muscular Atrophy; Cachexia; Sarcopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — * Blood sample (venous)
  * Muscle biopsy (vastus lateralis)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Muscle impaired elderly: Elderly scheduled for hip/knee/back surgery with III-IV ASA score, low grip strength and high scoring for sarcopenia
  Interventions: Other: In vitro analyse
- Lung cancer cachexia: Non-small cell lung cancer patients stage III with reported cachexia
  Interventions: Other: In vitro analyse
- Controls: Elderly scheduled for hip/knee/back surgery without any recorded muscle defects, I-II ASA score, average or high grip strength, low scoring for sarcopenia.
  Interventions: Other: In vitro analyse

INTERVENTIONS:
Other: In vitro analyse — In vitro analysis on isolated mesoangioblasts obtained from muscle biopsies

SUMMARY:
The goal of this clinical trial is to compare the quality of mesoangioblasts isolated from various patient groups suffering from muscle atrophy. This study includes cancer cachexia and muscle-impaired elderly and a control group of the same age.

The quality will be defined on these following outcomes:

* The number and distribution of the mesoangioblasts in a muscle biopsy to define if there are sufficient mesoangioblasts to start a culture.
* The proliferation capacity to define if we can culture them the numbers required for systemic treatment.
* The myogenic capacity to define if the mesoangioblasts are sufficiently capable to generate muscle fibres.

Participants will:

* Undergo a muscle biopsy (needle biopsy or rest material from surgery, ~50mg)
* Donate blood (~20 ml)
* Fill in SARC-F questionnaire (evaluate sarcopenia score)
* Fill in SQUASH questionnaire (evaluate physical activity of previous week) Researchers will compare groups (muscle-impaired elderly vs control; cancer cachexia vs control) to see if there is a difference regarding quality. These results will define the potential of autologous mesoangioblast therapy within these groups.

DETAILED DESCRIPTION:
No effective treatment is available for the loss of muscle tissue in non-genetic muscle diseases such as (cancer) cachexia and sarcopenia. Such a treatment would improve the quality of life, therapy success, and independency of these patients. The administration of healthy autologous muscle stem cells, called mesoangioblasts, that lead to muscle regeneration and increased muscle mass and function could be a novel therapeutic strategy to achieve this. A prerequisite is that the therapeutic potential of these mesoangioblasts is sufficient. Therefore, the main aim of this study is to assess this potential for mesoangioblasts of patients with lung cancer cachexia and with sarcopenia and determine the effect the cancer or age might have on the therapeutic potential.

This study is part of a larger project, called Generate Your Muscle (GYM), which aims to develop and commercially produce a stem cell therapy for recovery of muscle mass and strength in patients with genetic and non-genetic muscle disease and muscle breakdown. This will be achieved by administering large numbers of autologous mesoangioblasts (MABs) as an Advanced Therapy Medicinal Product (asCTMP) in the arteries, which will migrate to the damaged muscle, thereby restoring muscle mass and function. This strategy can only be successful for patients suffering from cachexia or sarcopenia, if these patients have enough mesoangioblasts, if these MABs can proliferate into the numbers requested for systemic treatment, if the energy capacity of the MABs is sufficient and if these mesoangioblasts still have a high myogenic potential. The aim of this study is to determine these parameters for patients with cancer cachexia or sarcopenia, as we know that they can be affected by the underlying condition. They will be compared to age-matched controls. If positive, the MABs will qualify as asCTMP for a clinical trial in a follow-up study.

ELIGIBILITY:
Inclusion Criteria:

Lung cancer cachexia:

* Diagnosed with NSCLC, stage III-IV
* Diagnosed with cachexia (>5% unintentional body weight loss in past six months, >2% body weight loss with BMI <20, or skeletal muscle index for males <7.26 kg/m2; females <5.45 kg/m2)
* Age 50-60 or 60-70
* Written informed consent

Patient group: MIE

* Scheduled for total hip, knee, or back surgery
* Age 60-70 or 70-80 year
* Written informed consent

Controls

* Patients with scheduled knee-, hip-, and back surgery
* Age 50-60, 60-70, and 70-80 year
* Age and sex-matched to patient groups
* Written informed consent

Exclusion Criteria:

* No filled-in IC
* Suffering from a muscular dystrophy or other disease known to affect muscle morphology or function
* Have a weekly alcohol intake of ≥ 35 units (men) or ≥ 24 units (women)
* Ongoing participation in other intervention clinical trials
* Major surgery of the muscle within 4 weeks of the visit unrelated to the study
* Patients unable and/or unwilling to comply with treatment and study instructions
* Any other factor that in the opinion of the investigator excludes the patient from the study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two study populations are included in this study. The Muscle Impaired Elderly (MIE) are considered elderly who struggle with muscle weakness. MIE is used as a substitute group for sarcopenia as their muscle weakness and daily impairments are confirmed, but confirmation via medical imaging lacks. Sarcopenia is multifactorial and the balance between nutrition and activity is disturbed.
  Cachexia is defined as an ongoing loss of skeletal muscle mass due to an illness that cannot be reversed by conventional nutrition and/or exercise. Lung cancer cachexia is a group where non-small cell lung cancer is confirmed along with non-intentional weight loss.
  Both groups will be compared to a Control group consisting of eldery undergoing knee/hip/back surgery but are otherwise considered healthy.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Number of mesoangioblasts ex vivo isolated from muscle biopsy | 1 day
  The number of mesoangioblasts obtained from a muscle biopsy. Once cells reached >80% confluency in a culture dish, FACS analysis will determine the amount of mesoangioblasts obtained.
Proliferation capacity of mesoangioblasts in vitro | 1 day
  The proliferation capacity to define whether we can culture them in the numbers required for systemic treatment. Doubling time will be assessed 3 separate instances with a hemocytometer. Population doubling level = 3.32 (log viable cells at harvest - log seeded cells)
Myogenic capacity of mesoangioblasts in vitro | 1 day
  The myogenic capacity to define if the mesoangioblasts are sufficiently capable to generate muscle fibres. Myogenic capacity is calculated as the number of nuclei in MF20-positive fibers divided by total number of nuclei per field.
Distribution of mesoangioblasts in a muscle biopsy | 1 day
  The number of mesoangioblasts in a muscle biopsy. Histochemistry will reveal the location of the pericyte-like mesoangioblasts surrounding the blood vessels when stained for pericyte marker NG2 proteoglycan.

SECONDARY OUTCOMES:
Homing potential of mesoangioblasts in vitro | 1 day
  The homing potential of the mesoangioblasts in these patients by characterizing inflammatory parameters via qPCR. Muscle damage reflected by inflammation is essential for the migration and engraftment of mesoangioblasts in the affected muscles. Differences in gene expression levels of cytokine IL6 and cytokine mediator HMGB1 in the groups MIE and Lung cancer patients vs Controls will be determined.
ATP production of mesoangioblasts in vitro | 1 day
  ATP production as a marker for metabolic health will be determined via the CellTiterGlo assay. Luminescence (Relative Light Unit) corrected for DNA content per well determines the ATP production.
Difference in myogenic potential of mesoangioblasts and satellite cells in vitro | 1 day
  Differences in myogenic potential between mesoangioblasts and satellite cells with respect due cachexia and sarcopenia. Myogenic capacity is calculated as the number of nuclei in MF20-positive fibers divided by total number of nuclei per field.